CLINICAL TRIAL: NCT06900842
Title: Chronic Pain in Mastectomy Patients; The Difference Between Pectoral Nerve Block (PECS I-II) and Erector Spinal Plane (ESP) Block
Brief Title: Chronic Pain in Post-Mastectomy Patients; The Difference Between Pectoral Nerve (PECS I-II) and Erector Spinal Plane (ESP) Blocks
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nurefsan Sadikoglu, Specialist in Anesthesiology, Hacettepe University
Other Study IDs: 2024/09-07 (KA-23086)
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Surgery; Postoperative Pain, Acute; Postoperative Pain, Chronic; Post-mastectomy Pain Syndrome; Regional Anesthesia; Pectoral Nerve (PECS) Block; Erector Spine Plane Block; Neuropathic Pain; Mastectomy; Quality of Life (QOL)
Keywords: breast cancer; Postoperative Pain; Chronic Pain; PECS I-II Block; Erector Spinae Plane Block; ESP Block; Chronic Pain Prevention; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings; Neuralgia; Breast Neoplasms; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PECS I-II Block Group: This group includes patients who received an ultrasound-guided pectoral nerve block (PECS I-II) before undergoing modified radical mastectomy (MRM). PECS I involved the injection of 10 mL of 0.25% bupivacaine between the pectoralis major and minor muscles. PECS II involved the injection of 20 mL of 0.25% bupivacaine between the pectoralis minor and serratus anterior muscles. The block was applied preoperatively at the discretion of the responsible anesthesiologist, independently from the study protocol. Postoperative pain scores, opioid requirements, and chronic pain development were evaluated.
- ESP Block Group: This group includes patients who received an ultrasound-guided erector spinae plane (ESP) block before undergoing modified radical mastectomy (MRM). The block was administered at the T4-T5 level, with 20-30 mL of 0.25% bupivacaine injected between the erector spinae muscle and the transverse process. The procedure was performed in the lateral decubitus position and verified via hydrodissection. The decision to perform this block was made independently by the anesthesiologist. Pain scores and analgesic use were tracked to assess the block's effect on acute and chronic postoperative pain.

SUMMARY:
This study looks at two types of injections (called PECS and ESP blocks) to see which one works better for reducing pain after breast cancer surgery (mastectomy).

The main question it asks is: Which block is better at reducing pain after surgery - PECS or ESP? Women who had this surgery and received one of the two blocks were followed for three months. We looked at how much pain they felt, how much pain medication they needed, and whether they still had pain months later.

The results showed that both blocks helped with pain right after surgery. The ESP block lasted a little longer at first, but in general, both groups needed about the same amount of pain medicine. Three months later, about half of the patients still had some pain - especially those who had more extensive surgery or had nerve pain early on. There was no big difference between the two blocks when it came to long-term pain.

DETAILED DESCRIPTION:
Despite advancements in breast cancer treatment, chronic postoperative pain-known as post-mastectomy pain syndrome (PMPS)-remains a common complication, with reported rates between 40-50%. It is typically neuropathic in nature and linked to factors such as axillary lymph node dissection, radiotherapy, and high levels of acute postoperative pain. Younger patients are at higher risk, and early neuropathic symptoms may predict long-term pain.

Regional anesthesia techniques, including PECS and erector spinae plane (ESP) blocks, are widely used to improve perioperative pain control and potentially reduce the incidence of chronic pain. These techniques are considered effective and low-risk adjuncts to general anesthesia.

This prospective observational study compares the impact of PECS I-II and ESP blocks on chronic pain development in patients undergoing modified radical mastectomy (MRM). The primary outcome is the incidence of pain at 3 months postoperatively (NRS ≥1). Secondary outcomes include acute pain scores, intraoperative fentanyl use, postoperative morphine requirements, and time to first analgesic. The study also explores associations between chronic pain and variables such as lymph node dissection, radiotherapy.

Findings aim to guide clinical practice in selecting regional anesthesia techniques that provide both immediate and long-term pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo modified radical mastectomy due to breast cancer
* Decision to perform PECS I-II or ESP block made independently from the study, as part of standard pain management
* Aged between 18 and 65 years
* American Society of Anesthesiologists (ASA) physical status classification I or II
* Female

Exclusion Criteria:

* Inability to perform the block (e.g., coagulation disorder, allergy to local anesthetics, infection at the injection site)
* Obesity (Body Mass Index > 35 kg/m²)
* Pre-existing neurological deficits
* Younger than 18 or older than 65 years
* ASA physical status classification III or IV
* Refusal to give informed consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study did not consider self-identified gender. Only individuals assigned female at birth were included.
Study Population: Study participants will be selected from female patients aged 18 to 65 years who are scheduled to undergo elective modified radical mastectomy for breast cancer at Hacettepe University Medical Faculty, Department of General Surgery. All participants must be classified as ASA physical status I or II and have received either a PECS I-II or ESP block as part of their routine pain management. Patients with significant comorbidities, pre-existing neurological deficits, or contraindications to regional anesthesia will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Chronic Postoperative Pain (NRS ≥1) | 3 months after surgery
  The presence of chronic pain will be evaluated at 3 months postoperatively using the Numeric Rating Scale (NRS). Patients reporting a score of ≥1 will be considered to have chronic postoperative pain. This measure aims to assess the long-term effectiveness of PECS I-II and ESP blocks in reducing chronic pain following mastectomy.

SECONDARY OUTCOMES:
Postoperative Acute Pain Scores (NRS) | At 20 minutes, 6 hours, and 24 hours after surgery
  Pain intensity will be measured using the Numeric Rating Scale (0-10). Scores will be compared between the PECS and ESP groups to evaluate differences in early postoperative pain control.
Total Postoperative Opioid Consumption (Morphine, mg) | Within 24 hours after surgery
  The total amount of intravenous morphine consumed via patient-controlled analgesia (PCA) pump will be recorded and compared between groups to assess analgesic requirements.
Time to First Analgesic Requirement | Within 24 hours after surgery
  The time interval from the end of surgery to the patient's first request for opioid analgesia will be recorded in minutes. This outcome reflects the duration of initial analgesia provided by the block.
Postoperative Quality of Life (SF-12 Score) | 3 months after surgery
  The SF-12 Health Survey will be used to assess the physical and mental components of quality of life. Results will be compared between groups and correlated with chronic pain presence.
Presence of Neuropathic Pain (DN4 Score > 4) | At 20 minutes, 6 hours, 24 hours, and 3 months after surgery
  In patients with NRS > 0, the DN4 (Douleur Neuropathic 4) questionnaire will be used to assess the presence of neuropathic pain. Scores > 4 indicate neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Documents will be shared upon request

REFERENCES:
- [Background] Banerjee S, Goswami R. GST profile expression study in some selected plants: in silico approach. Mol Cell Biochem. 2010 Mar;336(1-2):109-26. doi: 10.1007/s11010-010-0384-y. Epub 2010 Feb 5. PMID 20135200
- [Background] Carpenter JS, Andrykowski MA, Sloan P, Cunningham L, Cordova MJ, Studts JL, McGrath PC, Sloan D, Kenady DE. Postmastectomy/postlumpectomy pain in breast cancer survivors. J Clin Epidemiol. 1998 Dec;51(12):1285-92. doi: 10.1016/s0895-4356(98)00121-8. PMID 10086821
- [Background] Meijuan Y, Zhiyou P, Yuwen T, Ying F, Xinzhong C. A retrospective study of postmastectomy pain syndrome: incidence, characteristics, risk factors, and influence on quality of life. ScientificWorldJournal. 2013 Nov 27;2013:159732. doi: 10.1155/2013/159732. eCollection 2013. PMID 24379736
- [Background] Alves Nogueira Fabro E, Bergmann A, do Amaral E Silva B, Padula Ribeiro AC, de Souza Abrahao K, da Costa Leite Ferreira MG, de Almeida Dias R, Santos Thuler LC. Post-mastectomy pain syndrome: incidence and risks. Breast. 2012 Jun;21(3):321-5. doi: 10.1016/j.breast.2012.01.019. Epub 2012 Feb 27. PMID 22377590
- [Background] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Background] DeSantis CE, Ma J, Goding Sauer A, Newman LA, Jemal A. Breast cancer statistics, 2017, racial disparity in mortality by state. CA Cancer J Clin. 2017 Nov;67(6):439-448. doi: 10.3322/caac.21412. Epub 2017 Oct 3. PMID 28972651
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] Hanley MA, Jensen MP, Smith DG, Ehde DM, Edwards WT, Robinson LR. Preamputation pain and acute pain predict chronic pain after lower extremity amputation. J Pain. 2007 Feb;8(2):102-9. doi: 10.1016/j.jpain.2006.06.004. Epub 2006 Sep 1. PMID 16949876
- [Background] Tasmuth T, Kataja M, Blomqvist C, von Smitten K, Kalso E. Treatment-related factors predisposing to chronic pain in patients with breast cancer--a multivariate approach. Acta Oncol. 1997;36(6):625-30. doi: 10.3109/02841869709001326. PMID 9408154
- [Background] Miguel R, Kuhn AM, Shons AR, Dyches P, Ebert MD, Peltz ES, Nguyen K, Cox CE. The effect of sentinel node selective axillary lymphadenectomy on the incidence of postmastectomy pain syndrome. Cancer Control. 2001 Sep-Oct;8(5):427-30. doi: 10.1177/107327480100800506. PMID 11579339
- [Background] Steegers MA, Wolters B, Evers AW, Strobbe L, Wilder-Smith OH. Effect of axillary lymph node dissection on prevalence and intensity of chronic and phantom pain after breast cancer surgery. J Pain. 2008 Sep;9(9):813-22. doi: 10.1016/j.jpain.2008.04.001. Epub 2008 Jun 30. PMID 18585963
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Singh S, Chowdhary NK. Erector spinae plane block an effective block for post-operative analgesia in modified radical mastectomy. Indian J Anaesth. 2018 Feb;62(2):148-150. doi: 10.4103/ija.IJA_726_17. No abstract available. PMID 29491525
- [Background] Veiga M, Costa D, Brazao I. Erector spinae plane block for radical mastectomy: A new indication? Rev Esp Anestesiol Reanim (Engl Ed). 2018 Feb;65(2):112-115. doi: 10.1016/j.redar.2017.08.004. Epub 2017 Nov 2. English, Spanish. PMID 29102405
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- See also: Breast Cancer Facts & Figures 2019-2020 — https://www.cancer.org/content/dam/cancer-org/research/cancer-facts-and-statistics/breast-cancer-facts-and-figures/breast-cancer-facts-and-figures-2019-2020.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT06900842/Prot_SAP_000.pdf